

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

A phase I-II, open label study evaluating the safety and efficacy of alisertib and pembrolizumab in patients with Rb-deficient head and neck squamous cell carcinomas 2020-0210

| | 2000 X (1000 X |
|---|---|
| Study Chair: Faye Johnson | |
| <br>Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to find the highest tolerable dose of alisertib in combination with pembrolizumab when given to patients with head and neck squamous cell carcinomas (HNSCC). Researchers also want to learn if the combination has any effect on the disease.

The safety of this study drug combination will also be studied.

**This is an investigational study**. Alisertib is not FDA approved or commercially available. It is currently being used for research purposes only. Pembrolizumab is FDA approved and commercially available for the treatment of HNSCC. The study doctor can explain how the study drugs are designed to work.

Alisertib and pembrolizumab may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. You may not want to take part in this study

due to the availability of other treatments or an inability to visit MD Anderson for extra visits.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You may receive the study drugs for as long as the study doctor thinks it is in your best interest.

Alisertib will be provided at no cost to you during this study. You and/or you insurance provider will be responsible for the cost of pembrolizumab.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other FDA approved drugs, such as chemotherapy or immunotherapy (such as pembrolizumab). The study doctor can discuss these alternatives with you, along with their potential risks and benefits. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer. Talk to your study doctor about your choices before you decide if you will take part in this study.

#### 1. STUDY DETAILS

# **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be done within 22 days before your first dose of study drugs to help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an EKG to check your heart function.
- Blood (about 5-7 teaspoons) will be drawn for routine tests and to test for HIV (the AIDS virus), hepatitis B, and hepatitis C.
- Blood (about 3 tablespoons) will be drawn for biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drugs.
- You will have a CT scan or MRI to check the status of the disease.
- If you can become pregnant, blood (about 1-2 teaspoons) or urine will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

#### **Study Groups**

If you are found to be eligible to take part in this study, you will be assigned to a dose level of alisertib based on when you join this study. Up to 3 dose levels of alisertib will be tested. About 3-9 participants will be enrolled at each dose level. The first group of participants will receive the starting dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. There is a possibility that a lower dose level than the starting dose may also be tested, depending

on the results seen. This will continue until the highest tolerable dose of alisertib is found. This is called dose escalation.

As of March 2022, a recommended dose has been found. Additional patients will be enrolled to receive this dose of alisertib in combination with pembrolizumab. This is called dose expansion. Please note, the addition of alisertib to your treatment plan may delay and/or interrupt your treatment with pembrolizumab due to possible side effects from alisertib.

All participants will receive the same dose of pembrolizumab.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

#### Study Drug Administration

Each study cycle is 21 days.

You will receive pembrolizumab by vein over about 30 minutes on Day 1 of every cycle.

You will take alisertib tablets by mouth 2 times a day on Days 1-7 of each cycle. Each dose should be taken at about the same time each day at least 6 hours apart. Alisertib tablets should be swallowed whole with a full glass (about 8 ounces) of water.

If you cannot swallow whole tablets or if you have a feeding tube in place, you will be given a liquid version of alisertib. The liquid version must be given on an empty stomach, at least one hour before and two hours after food or drink except water.

If you miss or vomit a dose of alisertib, do not take a "make up" dose. Wait and take your next dose as scheduled.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

# **Study Visits**

## On Day 1 of every cycle:

- You will have a physical exam.
- Blood (about 5-7 teaspoons) will be drawn for routine tests.
- During Cycle 1 only, if you are one of the first 12 participants enrolled in the dose expansion part of the study, blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing before the dose and then 5 more times over the 10 hours after the dose. PK testing measures the amount of study drugs in the body at different time points.
- If you can become pregnant, blood (about 1-2 teaspoons) or urine will be collected for a pregnancy test.

# On Day 7 of Cycle 1:

- You will have a physical exam.
- Blood (about 4-6 teaspoons) will be drawn for routine tests.

- If you are one of the first 12 participants enrolled in the dose expansion part of the study, blood (about 1 teaspoon each time) will be drawn for PK testing before the dose and then 5 more times over the 10 hours after the dose.
- Every 2 cycles, you will have an MRI or CT scan to check the status of the disease and blood (about 3 tablespoons) will be drawn for biomarker testing.

# **End of Dosing Visit**

At the next clinic visit after your last dose of study drugs:

- You will have a physical exam.
- Blood (about 4-6 teaspoon) will be drawn for routine tests.
- You will have an EKG.

# Follow up

Every 2-3 months after your last dose of study drugs, the study staff will either review your medical record or call you to find out how you are doing and if you have started any new medications. Each call should last about 5-10 minutes. This follow-up will continue for up to 3 years.

# **Other Information**

- The use of live vaccines (such as the flu vaccine or the measles, mumps, rubella [MMR] vaccine) and close contact with those who have received live vaccines should be avoided while taking the study drug.
- You must avoid grapefruit juice and grapefruit-containing products while taking the study drug.
- You must limit the use of alcohol while enrolled in this study. Do not have more than 1 standard unit of alcohol per day during the study and for 30 days from the last dose of alisertib. A standard unit of alcohol is defined as a 12 ounce beer (350 mL), 1½ ounces (45 mL) of 80-proof alcohol, or one 6-ounce (175 mL) glass of wine.
- Until you know how the study drugs affect you, you should not drive or engage in any hazardous activities (such as operating heavy machinery). You should also have a family member or caregiver drive you or check in on you while you are receiving the study drugs (as alisertib may cause sleepiness, memory loss, and/or confusion).

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

Pembrolizumab and alisertib may commonly cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue.
   You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Pembrolizumab Side Effects

# Common (occurring in more than 20% of patients)

- fatigue
- fever
- skin rash and/or itching
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- high blood sugar (possible diabetes)
- high blood levels of fat (possible heart disease and/or stroke)
- loss of appetite
- nausea
- constipation
- diarrhea
- abdominal pain

- low blood cell counts (red, white, platelets)
- abnormal liver test (possible liver damage)
- pain
- abnormal kidney test (possible kidney damage)
- cough
- difficulty breathing

# Occasional (occurring in 3-20% of patients)

- swelling (face/arm/leg)
- inflammation of the tissue around the heart (possible chest pain)
- irregular heartbeat
- headache
- confusion
- patches of skin color loss
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- overactive thyroid gland (possible weight loss, diarrhea, mood swings, difficulty sleeping, heart rate changes, and/or sweating)
- low blood sugar
- weight loss
- fluid in the abdomen
- blood in the urine
- vomiting
- abnormal liver test (possible yellowing of the skin and/or eyes)

- weakness
- nerve damage (possible numbness, pain, and/or loss of motor function)
- difficulty breathing (possibly due to lung inflammation)
- flu-like symptoms
- infusion reaction (possible dizziness, low blood pressure, nausea, pain, and/or difficulty breathing)

# Frequency Unknown

- heart failure
- heart attack
- build-up of fluid around the heart (possible heart failure)
- abnormal connections or passageways between organs or vessels
- bleeding in the rectum and/or uterus
- blockage in the lung (possible pain and/or shortness of breath)
- nosebleed
- coughing up blood

# Rare but serious (occurring in fewer than 3% of patients)

- low blood pressure (possible dizziness/fainting)
- heart inflammation
- build-up of fluid in the tissue around the heart
- blood vessel inflammation (possible bleeding, skin rash, numbness/weakness, fever, weight loss, fatigue, and/or bruising, depending on where the inflammation occurs)
- seizure
- immune system damage to the nervous system (causing muscle weakness, numbness and/or paralysis)
- spinal cord inflammation (possible pain, weakness, loss of feeling or movement, and/or paralysis)
- brain inflammation (possible paralysis and/or coma)
- shedding, scaling and/or inflammation of the skin (possible fatal loss of bodily fluids)
- large skin blisters
- very severe blistering skin disease (loss of large portion of skin

- low hormone blood levels (possible weakness, bone changes, and/or cramping)
- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- pituitary gland inflammation (possible headaches)
- inflammation of the thyroid gland (possible tenderness in the neck)
- diabetes requiring insulin
- severe high blood sugar due to uncontrolled diabetes
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- low pancreatic enzyme level (possible bloating, gas, abdominal discomfort, diarrhea, oily stool, and/or weight loss)
- inflammation of the pancreas (possible abdominal pain)
- inflammation of the stomach (possible belly

- inflammation inside the eye (possible vision problems)
- kidney inflammation (possible kidney damage/failure)
- kidney failure
- inflammation of an eye nerve (possible vision loss, loss of color vision, pain when moving your eyes, and/or loss of peripheral vision in one or both eyes)
- build-up of fluid around the lungs
- immune response that causes the body to attack itself (possible organ damage)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- immune response (causing muscle weakness)
- immune system reaction (possible fever, jaundice, liver/spleen enlargement, irritability, and/or seizures)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)

pale or yellow skin, dark urine, or fever.

If you have a solid tumor type and you have an organ transplant, pembrolizumab may increase your risk for the transplant to be rejected by your body.

Pembrolizumab works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue. These side effects can affect more than one of your normal organs and tissues at the same time.

## **Alisertib Side Effects**

# Common (occurring in more than 20% of patients)

| <ul> <li>sleepiness</li> <li>fatigue</li> <li>fever</li> <li>hair loss (partial or total)</li> </ul> | <ul> <li>mouth blisters/sores<br/>(possible difficulty<br/>swallowing)</li> <li>diarrhea</li> </ul> | <ul> <li>nausea/vomiting</li> <li>loss of appetite</li> <li>low blood cell counts<br/>(red/platelets/white)</li> </ul> |
|---|---|---|
|---|---|---|

# Occasional (occurring in 3-20% of patients)

- high blood pressure
- low blood pressure (possible dizziness/fainting)
- swelling (arm/leg)
- abnormal heartbeat
- chills
- headache
- dizziness
- confusion
- weakness
- anxiety or depression
- difficulty sleeping
- skin rash
- itching
- hand-foot syndrome (palms of hands/soles of feet having pain, swelling, and blistering)
- dry skin
- high blood sugar (possible diabetes)

- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- constipation
- dehydration
- weight loss
- abdominal swelling
- upset stomach
- gas
- hemorrhoids
- dry mouth
- difficulty swallowing

- abnormal taste
- voice problems (possible hoarseness and difficulty speaking)
- increased risk of bleeding
- abnormal liver tests (possible liver damage)
- muscle spasms
- pain
- blurry vision
- fluid around the lung or abdomen
- cough
- difficulty breathing
- infection
- lymph node swelling

# Rare but serious (occurring in fewer than 3% of patients)

- severe heart problems
- heart attack
- memory loss
- nerve damage (possible numbness, tingling, and pain)
- shock
- •

- severe blisters
- sweating
- loss of balance (possible falling)
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- blood clot (usually in the legs)
- destruction of red blood cells

- liver damage due to blood clots
- abnormal kidney function
- breakdown of muscle tissue (possible kidney failure)
- failure of multiple organs
- body-wide inflammation
- hearing loss
- · ringing in the ears

Alisertib may rarely cause you to develop another type of cancer (such as leukemia, a type of blood cancer).

You should use caution while driving, operating dangerous machinery, or performing any other task requiring full alertness and/or coordination. If you experience sleepiness, confusion, or memory loss, avoid performing these tasks entirely.

A safety review was completed after the first 12 patients received the study drug. Three (3) patients died during active treatment. One of these fatalities was due to the patient's cancer rapidly worsening. The others experienced complications related to the blood, heart and lungs; specifically destruction of red blood cells, abnormal blood clotting in small blood vessels, heart attack, and respiratory failure. It is not known if these were associated with the patients' cancer, their other medical conditions, or side effects due to the study drug(s). You will be closely monitored for any side effects while you are on study.

**Liquid alisertib** contains propylene glycol and polyethylene glycol 400, which are oily, colorless inactive ingredients. The concentration of these ingredients is within the range of levels used in FDA approved drug products and is generally considered safe for use in liquid drugs.

When large amounts of propylene glycol are swallowed, it may cause an increased risk of metabolic acidosis. Metabolic acidosis is a chemical imbalance which may cause convulsions, nausea, vomiting, headache, and loss of consciousness and slowing of the heart and breathing rate.

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study

doctor.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**.

This study may involve unpredictable risks to the participants.

# **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study and for 120 days after your last dose of study drugs, if you are sexually active.

If you can become pregnant or father a child, you must use 1 highly effective method of birth control (such as birth control pills, implants, and injections) and 1 barrier method (condom, diaphragm, or cervical cap).

Males: Do not donate sperm while on study and for at least 120 days after the last dose of study drugs. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy. If your partner/spouse becomes pregnant while you are on this study, the sponsor would like to collect information about the pregnancy. The study sponsor's contact information will be made available so that, if you and your partner wish to, you can share information about the outcome of the pregnancy with the sponsor. If you and/or your partner choose not to share this information, it will not result in any penalty or loss of benefits to which you are otherwise entitled.

Females: Do not donate eggs while on study and for at least 120 days after the last dose of study drugs. If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. The sponsor will ask for information about the pregnancy.

Getting pregnant will result in your removal from this study.

#### OPTIONAL PROCEDURES FOR THE STUDY

**Optional Procedure #1:** If you are in the dose expansion part of the study and you agree, you will have a tumor biopsy for biomarker testing at screening and then about 6

weeks after your first dose of study drugs. The type of biopsy you have will depend on where the tumor is located. This will be discussed with you.

There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

# **Optional Procedure Risks**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

#### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have a biopsy at screening and then about 6 weeks after your first dose of study drugs?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Puma Biotechnology for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result

from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Faye Johnson, at 713-792-6363) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. It may be dangerous to suddenly stop study treatment, and the study doctor can discuss ways to safely withdraw. If you withdraw from this study, you can still choose to be treated at MD Anderson.

The study staff may ask if they can continue collecting the results of routine care from your medical record.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Puma Biotechnology, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will not contact you to let you know what they have found.

- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Puma Biotechnology.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

## **Future Research Data**

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and Puma Biotechnology, and/or shared with

other researchers and/or institutions for use in future research.

# **Samples**

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples

#### **Genetic Research**

Samples collected from you as part of this study may be used for genetic research, which may include whole exome sequencing. Whole exome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment.

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

# **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Puma Biotechnology, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
  - Any future sponsors and/or licensees of the study technology.
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At

most, the Web site will include a summary of the results. You can search this Web site at any time.

## **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT **WITNESS TO CONSENT** I was present during the explanation of the research to be performed under this protocol. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. PRINTED NAME OF WITNESS TO THE VERBAL CONSENT PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her authorized representative, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE PRINTED NAME OF PERSON OBTAINING CONSENT **TRANSLATOR** I have translated the above informed consent as written (without additions or and assisted the people subtractions) into (Name of Language) obtaining and providing consent by translating all questions and responses during the consent process for this participant. NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DATE Please check here if the translator was a member of the research team. (If checked, a witness, other

than the translator, must sign the witness line.)